CLINICAL TRIAL: NCT04622319
Title: A Phase 3, Multicenter, Randomized, Open-Label, Active-Controlled Study of Trastuzumab Deruxtecan (T-DXd) Versus Trastuzumab Emtansine (T-DM1) in Participants With High-Risk HER2-Positive Primary Breast Cancer Who Have Residual Invasive Disease in Breast or Axillary Lymph Nodes Following Neoadjuvant Therapy (DESTINY-Breast05)
Brief Title: A Study of Trastuzumab Deruxtecan (T-DXd) Versus Trastuzumab Emtansine (T-DM1) in High-risk HER2-positive Participants With Residual Invasive Breast Cancer Following Neoadjuvant Therapy (DESTINY-Breast05)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry); NSABP Foundation Inc (Network); GBG Forschungs GmbH (Other); Spanish Breast Cancer Research Group (SOLTI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-U305; 2020-003982-20 (EudraCT Number); DESTINY-Breast05 (Other: Daiichi Sankyo and AstraZeneca); NSABP B-60 (Other: National Surgical Adjuvant Breast and Bowel Project (NSABP)); GBG-103 (Other: German Breast Group (GBG)); SOLTI-2001 (Other: Spanish Breast Cancer Research Group (SOLTI))
Record Dates: First submitted 2020-11-02; First posted 2020-11-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: HER2-Positive Primary Breast Cancer; Residual Invasive Breast Cancer
Keywords: HER2-Positive Primary Breast Cancer; Residual Invasive Breast Cancer; Trastuzumab Deruxtecan; Trastuzumab Emtansine
MeSH Terms: interventions — trastuzumab deruxtecan; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trastuzumab deruxtecan (T-DXd) (Experimental): Participants who will be randomized to receive trastuzumab deruxtecan (T-DXd) at a starting dose of 5.4 mg/kg.
  Interventions: Drug: DS-8201a
- Trastuzumab ematansine (T-DM1) (Active Comparator): Participants who will be randomized to receive trastuzumab ematansine (T-DM1) at a starting dose of 3.6 mg/kg.
  Interventions: Drug: T-DM1

INTERVENTIONS:
Drug: DS-8201a — Administered initially as an intravenous (IV) infusion at a dose of 5.4 mg/kg on Day 1 of each 21-day cycle
  Other Names: Trastuzumab deruxtecan (T-DXd)
  Arms: Trastuzumab deruxtecan (T-DXd)
Drug: T-DM1 — Administered initially as an intravenous (IV) infusion at a dose of 3.6 mg/kg on Day 1 of each 21-day cycle
  Other Names: Trastuzumab emtansine (T-DM1)
  Arms: Trastuzumab ematansine (T-DM1)

SUMMARY:
Patients with HER2-positive primary breast cancer (BC) who do not achieve complete response after appropriate neoadjuvant therapy are at higher risk of disease recurrence. More effective treatment options are needed for this patient population. This study will examine the efficacy and safety of trastuzumab deruxtecan (T-DXd) compared with trastuzumab emtansine (T-DM1) in high-risk patients with residual invasive breast cancer following neoadjuvant therapy.

DETAILED DESCRIPTION:
This study will examine trastuzumab deruxtecan (T-DXd) versus trastuzumab emtansine (T-DM1) in patients with HER2-positive primary BC who have residual invasive disease in breast or axillary lymph nodes with higher risk of recurrence, which includes patients who were inoperable at disease presentation or had pathological node-positive status after neoadjuvant therapy.

The primary objective is to compare invasive disease-free survival (IDFS) between T-DXd and T-DM1 treatment arms in this population. The key secondary objective of the study is to evaluate disease-free survival (DFS).

ELIGIBILITY:
Key Inclusion Criteria:

* Adults ≥18 years old (local regulatory requirements will apply if the legal age of consent for study participation is >18 years old).
* Pathologically documented HER2-positive breast cancer (BC):

  * HER2-positive expression defined as an immunohistochemistry (IHC) score of 3+ and/or positive by in situ hybridization (ISH) confirmed prior to study randomization.
* Histologically confirmed invasive breast carcinoma.
* Clinical stage at disease presentation: T1-4, N0-3, M0; patients presenting with T1N0 tumors are not eligible.
* Pathologic evidence of residual invasive carcinoma in the breast and/or axillary lymph nodes following completion of neoadjuvant therapy meeting one of the following high-risk criteria:

  * Inoperable breast cancer at presentation (prior to neoadjuvant therapy), defined as clinical stages T4, N0-3, M0 or T1-3, N2-3, M0.
  * Operable at presentation, defined as clinical stages T1-3,N0-1,M0, with axillary node positive disease (ypN1-3) following neoadjuvant therapy.
* Completion of neoadjuvant systemic therapy, including taxane-based chemotherapy and HER2-directed treatment prior to surgery.

  * Systemic therapy must consist of at least 6 cycles of neoadjuvant therapy with a total duration of at least 16 weeks, including at least 9 weeks of trastuzumab (± pertuzumab) and at least 9 weeks of taxane-based chemotherapy to be completed prior to surgery. Patients may have received an anthracycline as part of neoadjuvant therapy in addition to taxane chemotherapy.
* Adequate excision as confirmed per medical records: surgical removal of all clinically evident disease in the breast and axillary lymph nodes.
* An interval of no more than 12 weeks between the date of last surgery and the date of randomization.
* Known hormone receptor (HR) status, per local laboratory assessment, as defined by ASCO-CAP guidelines (≥1%): HR positive status defined by either positive estrogen receptor (ER) and/or positive progesterone receptor (PR).

status. HR-negative status defined by both known negative ER and known negative PR.

* Left ventricular ejection fraction (LVEF) ≥50% within 28 days prior to randomization.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at Screening.
* Has adequate organ function within 14 days before randomization.

Key Exclusion Criteria:

* Stage IV (metastatic) BC.
* History of any prior (ipsi- or contralateral) breast cancer except lobular carcinoma in situ (LCIS).
* Evidence of clinically evident gross residual or recurrent disease following neoadjuvant therapy and surgery.
* Prior treatment with T-DXd, T-DM1 or other anti-HER2 antibody-drug conjugate (ADC) or prior enrollment in a clinical study of T-DXd (regardless of treatment arm)
* History of exposure to the following cumulative doses of anthracyclines:

  * Doxorubicin > 240 mg/m^2
  * Epirubicin or Liposomal Doxorubicin-Hydrochloride > 480 mg/m^2
  * For other anthracyclines, exposure equivalent to doxorubicin > 240 mg/m^2
* History of other malignancy within the last 5 years except for appropriately treated CIS of the cervix, nonmelanoma skin carcinoma, Stage I melanoma skin carcinoma, Stage I uterine cancer, or other appropriately treated non-breast malignancies with an outcome similar to those mentioned above.
* History of (noninfectious) interstitial lung disease (ILD)/pneumonitis that required steroids and/or has ILD/pneumonitis noted on computed tomography (CT) scan of the chest at Screening (asymptomatic interstitial changes confined to recent radiation therapy fields are not excluded).
* Known pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (eg, pulmonary emboli within three months prior to randomization, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease).
* Any autoimmune, connective tissue or inflammatory disorders (eg, Rheumatoid arthritis, Sjogren's, sarcoidosis, etc) where there is documented or a suspicion of pulmonary involvement or pneumonectomy at the time of screening.
* Medical history of myocardial infarction (MI) within 6 months before randomization, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV), troponin levels consistent with MI as defined according to the manufacturer 28 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (IDFS) in Participants Who Were Administered Trastuzumab Deruxtecan (T-DXd) Compared With Trastuzumab Emtansine (T-DM1) Treatment | Randomization to date of invasive local, axillary or distant recurrence, invasive contralateral breast cancer or death from any cause (whichever occurs first), up to approximately 57 months postdose

SECONDARY OUTCOMES:
Disease-free Survival (DFS) in Participants Who Were Administered Trastuzumab Deruxtecan (T-DXd) Compared With Trastuzumab Emtansine (T-DM1) Treatment | Randomization to date of the first occurrence of an IDFS event including second primary non-breast cancer event or contralateral or ipsilateral ductal carcinoma in situ (whichever occurs first), up to approximately 81 months postdose
Overall Survival (OS) in Participants Who Were Administered Trastuzumab Deruxtecan (T-DXd) Compared With Trastuzumab Emtansine (T-DM1) Treatment | Randomization to date of death from any cause, up to approximately 81 months postdose
Distant Recurrence-free Interval (DRFI) in Participants Who Were Administered Trastuzumab Deruxtecan (T-DXd) Compared With Trastuzumab Emtansine (T-DM1) Treatment | Randomization to date of distant recurrence, up to approximately 81 months postdose
Brain Metastases-free Interval (BMFI) in Participants Who Were Administered Trastuzumab Deruxtecan (T-DXd) Compared With Trastuzumab Emtansine (T-DM1) Treatment | Randomization to date of brain metastasis, up to approximately 81 months postdose
Percentage of Treatment-emergent Adverse Events in Participants Who Were Administered Trastuzumab Deruxtecan (T-DXd) Compared With Trastuzumab Emtansine (T-DM1) Treatment | Baseline up to approximately 81 months postdose
Serum Concentrations of Trastuzumab Deruxtecan (T-DXd), total anti-HER2 antibody, and Active Metabolite MAAA-1181a | Pre-dose on Day 1 of Cycles 1, 4 and 10 and within 15 minutes post-dose on Day 1 of Cycles 1 and 4 (each cycle is 21 days)
Percentage of Participants Positive for Treatment-emergent Anti-drug Antibodies (ADAs) in Participants Who Were Administered Trastuzumab Deruxtecan (T-DXd) | Baseline up to approximately 81 months postdose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (480):
- United States (125):
  - The Oncology Institute of Hope & Innovation, Anaheim, California
  - Kaiser Permanente, Anaheim, California
  - Kaiser Permanente, Baldwin Park, California
  - Kaiser Permanente, Bellflower, California
  - Kaiser Permanente, Fontana, California
  - Orange Coast Blood and Cancer Care, Fountain Valley, California
  - Kaiser Permanente, Harbor City, California
  - Kaiser Permanente, Irvine, California
  - Long Beach Memorial TCI, Long Beach, California
  - Kaiser Permanente, Los Angeles, California
  - Kaiser Permanente, Ontario, California
  - Kaiser Permanente, Panorama City, California
  - Kaiser Permanente, Riverside, California
  - Kaiser Permanente, San Diego, California
  - Kaiser Permanente, San Marcos, California
  - Kaiser Permanente, West Los Angeles, California
  - Kaiser Permanente, Woodland Hills, California
  - SCRI FCS North- Altamonte, Altamonte Springs, Florida
  - SCRI FCS South- Bonita, Bonita Springs, Florida
  - SCRI FCS North- Brandon Cancer Center, Brandon, Florida
  - SCRI FCS South- North Fort Myers, Cape Coral, Florida
  - SCRI FCS North- Mease/Clearwater, Clearwater, Florida
  - SCRI FCS South, Fort Myers, Florida
  - SCRI FCS South- Colonial, Fort Myers, Florida
  - SCRI FCS South- Gladiolus, Fort Myers, Florida
  - SCRI FCS North- Gainesville Cancer Center, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - SCRI FCS North- Villages East, Lady Lake, Florida
  - SCRI FCS South- Lakewood Ranch, Lakewood Rch, Florida
  - SCRI FCS North- Largo/Highland, Largo, Florida
  - SCRI FCS North- Lecanto, Lecanto, Florida
  - SCRI FCS South- Naples West, Naples, Florida
  - SCRI FCS South- Naples/Goodlette, Naples, Florida
  - SCRI FCS North- New Port Richey, New Port Richey, Florida
  - SCRI FCS North- Ocala, Ocala, Florida
  - Orlando Health, Ocoee, Florida
  - SCRI FCS North- Orange City, Orange City, Florida
  - Orlando Health, Orlando, Florida
  - SCRI FCS North- Orlando Downtown, Orlando, Florida
  - SCRI FCS South- Port Charlotte, Port Charlotte, Florida
  - SCRI FCS South- Sarasota-Cattleman, Sarasota, Florida
  - SCRI FCS South-Sarasota-Downtown, Sarasota, Florida
  - SCRI FCS North- Spring Hill, Spring Hill, Florida
  - SCRI FCS North- St. Anthony's/St. Petersburg, St. Petersburg, Florida
  - SCRI FCS North, St. Petersburg, Florida
  - SCRI FCS North- Tampa Cancer Center, Tampa, Florida
  - SCRI FCS North- Tavares, Tavares, Florida
  - SCRI FCS South- Venice Healthpark, Venice, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - SCRI FCS North- Winter Park, Winter Park, Florida
  - Elmhurst Memorial Hospital- Nancy W. Knowles Cancer Center, Elmhurst, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Edward Cancer Center Plainfield, Plainfield, Illinois
  - University of Kentucky, Markey Cancer Center, Clinical Research Organization, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - LSU Health Baton Rouge North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group-Medical Oncology, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - MedStar Franklin Square Medical Center-Harry and Jeanette Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Franklin Square Cancer Center at Loch Raven Campus, Baltimore, Maryland
  - Frederick Health-James M Stockman Cancer Center, Frederick, Maryland
  - Maryland Oncology Hematology, Silver Spring, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Montefiore Medical Center, The Bronx, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - UNC Cancer Care at Nash, Rocky Mount, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic - Hillcrest, Cleveland, Ohio
  - Cleveland Clinic-Fairview, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Cleveland Clinic South Pointe, Warrensville Heights, Ohio
  - UPMC Upper St. Clair, Bethel Park, Pennsylvania
  - UPMC Passavant Cranberry/North, Cranberry Township, Pennsylvania
  - UPMC Erie, Erie, Pennsylvania
  - AHN Cancer Inst at St Vincent, Erie, Pennsylvania
  - UPMC Arnold Palmer-Mt View, Greensburg, Pennsylvania
  - UPMC Pinnacle-Ortenzio Cancer Center, Harrisburg, Pennsylvania
  - UMPC Pinnacle Pharmacy, Harrisburg, Pennsylvania
  - AHN Cancer Insititute at Jefferson, Jefferson Hills, Pennsylvania
  - AHN Cancer Institute at Forbes, Monroeville, Pennsylvania
  - UPMC Monroeville, Monroeville, Pennsylvania
  - UPMC Arnold Palmer-Mt Pleasant, Mount Pleasant, Pennsylvania
  - UPMC Arnold Palmer-Norwin, N. Huntingdon, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Magee, Pittsburgh, Pennsylvania
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - AHN Cancer Inst at West Penn, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Passavant HOA, Pittsburgh, Pennsylvania
  - UPMC Passavant OHA, Pittsburgh, Pennsylvania
  - UPMC Uniontown, Uniontown, Pennsylvania
  - UPMC Washington, Washington, Pennsylvania
  - Reading Hospital, McGlinn Cancer Institute, West Reading, Pennsylvania
  - AHN Cancer Institute at Wexford, Wexford, Pennsylvania
  - UPMC Pinnacle-Memorial Cancer Center, York, Pennsylvania
  - SCRI TO Nashville- Franklin Tennessee Oncology, PLLC, Franklin, Tennessee
  - SCRI TO Nashville- Gallatin Tennessee Oncology, PLLC, Gallatin, Tennessee
  - SCRI TO Nashville- Hendersonville Tennessee Oncology, PLLC, Hendersonville, Tennessee
  - SCRI TO Nashville- Summit Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - SCRI TO Nashville- Lebanon Tennessee Oncology, PLLC, Lebanon, Tennessee
  - SCRI TO Nashville- St. Thomas Midtown Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology Nashville / Sarah Cannon, Nashville, Tennessee
  - SCRI TO Nashville- St. Thomas West Tennessee Oncology, PLLC, Nashville, Tennessee
  - SCRI TO Nashville- Skyline Tennessee Oncology, PLLC, Nashville, Tennessee
  - SCRI TO Nashville- Southern Hills Tennessee Oncology, PLLC, Nashville, Tennessee
  - SCRI TO Nashville- Smyrna Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Houston Methodist Baytown, Baytown, Texas
  - Houston Methodist, Houston, Texas
  - Houston Methodist Willowbrook, Houston, Texas
  - Houston Methodist West, Houston, Texas
  - Houston Methodist Clear Lake, Nassau Bay, Texas
  - Houston Methodist Sugarland, Sugar Land, Texas
  - Houston Methodist Woodlands, The Woodlands, Texas
  - Wellmont Medical Associates Oncology & Hematology, Bristol, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - MultiCare Cancer Center Aurburn, Auburn, Washington
  - MultiCare Regional Cancer Center - Gig Harbor, Gig Harbor, Washington
  - MultiCare Cancer Center Puyallup, Puyallup, Washington
  - MultiCare Institute for Research & Innovation, Spokane, Washington
  - MultiCare Cancer Center Tacoma, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
- Argentina (6):
  - Centro Oncologico Riojano Integral, Capital, La Rioja Province
  - Sanatorio Británico de Rosario, Rosario, Santa Fe Province
  - Instituto de Oncología de Rosario, Rosario, Santa Fe Province
  - COIBA, Buenos Aires
  - Instituto Alexander Fleming, Caba
  - CER San Juan, San Juan
- Australia (9):
  - Royal Adelaide Hospital, Adelaide
  - Chris O Brien Lifehouse, Camperdown
  - Monash Health, Clayton
  - Austin Hospital- Olivia Newto-John Cancer and Wellness Centre, Heidelberg
  - Peter MacCallum Cancer Centre, Melbourne
  - Breast Cancer Research Centre - WA, Nedlands
  - Genesis Care Northern Cancer, Saint Leonards
  - St John of God Hospital - Bendat Family Comprehensive Cancer Centre (BFCCC), Subiaco
  - Southern Medical Day Care Centre, Wollongong
- Belgium (8):
  - Antwerp University Hospital, Edegem, Antwerpen
  - UZ Gent, Ghent, O. VL.
  - Algemeen Ziekenhuis AZ Klina - Borstkliniek, Brasschaat
  - Institut Jules Bordet Brussels Belgium, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven - Campus Gasthuisberg, Leuven
  - CHU Liege, Liège
  - GZA Hospitals Campus Sint- Augustinus, Wilrijk
- Brazil (9):
  - Hospital Sirio-Libanes HSL - Centro de Oncologia - Brasilia, Brasília, Federal District
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Fundação Universidade de Caxias do Sul Instituto de Pesquisas em Saúde IPS-UCS, Caxias do Sul, Rio Grande do Sul
  - Hospital Sao Lucas PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII-Hospital de Cancer de Barretos, Barretos, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - INCA - Instituto Nacional do Cancer / Hospital do Cancer HCIII, Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo (ICESP), São Paulo
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - CIUSSSS de l'Est-de-l'Ile-de-Montréal - Installation Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM, Montreal, Quebec
  - Jewish General Hospital Segal Cancer Centre, Montreal, Quebec
  - McGill University Health Centre - Cedars Cancer Centre, Montreal, Quebec
  - CHU de Quebec - Hopital du Saint-Sacrement, Québec, Quebec
- Chile (3):
  - Hospital Clinico Universidad de Chile, Santiago, RM
  - Fundacion Arturo Lopez Perez, Santiago
  - SIM CRC, Temuco
- China (17):
  - Peking University Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Jilin University JLU - First Affiliated Hospital, Changchun
  - Sichuan University - West China Hospital, Chengdu
  - Chongqing Medical University - The First Affiliated Hospital, Chongqing
  - Union Hospital of Fujian Medical University, Fuzhou
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Guangdong Academy of Medical Science, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Second Affiliated Hospital of Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Nanchang University - The First Affiliated Hospital, Nanchang
  - Nanjing Medical University NMU - Jiangsu Province Hospital, Nanjing
  - Fudan University Cancer Hospital, Shanghai
  - The 4th Hospital of Heibei Medical University, Shijiazhuang
  - The First Affiliated Hospital of Xiamen University, Xiamen
- Czechia (2):
  - University Hospital Brno, Brno
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Soenderborg sygehus, Syddanmark
- France (21):
  - Clinique Tivoli Ducos - Centre dOncologie et de Radiotherapie a Bordeaux, Bordeaux, Gironde
  - Institut Claudius Regaud, Toulouse, Haute Garonne
  - CHR Metz-Thionville, Metz, Lorraine
  - Institut De Cancerologie De La Loire, Saint-Priest-en-Jarez, Pays de la Loire Region
  - Institut Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - CHD Vendee, La Roche-sur-Yon
  - Centre Hosp Univ de Grenoble CHUG, La Tronche
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - The Sel of Centre dOncologie de Gentilly, Nancy
  - Centre Antoine Lacassagne, Nice
  - Hospital St Louis, Paris
  - Hopital Georges Pompidou, Paris
  - IUC AP-HP. Sorbonne Université, Hôpital Tenon, Paris
  - CHU de Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes
  - Institut de cancerologie de l'ouest, Saint-Herblain
  - Strasbourg Europe Cancer Institute, Strasbourg
- Germany (81):
  - Gemeinschaftspraxis Dres. Halder / Bangerter, Augsburg
  - Cahrité Campus Mitte, Berlin
  - Praxis Dr. med. J. Schilling, Berlin
  - MediOnko-Institut GbR, Praxisklinik Krebsheilkunde, Berlin
  - DRK Kliniken Berlin Köpenick, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Onkologische Schwerpunktpraxis, Berlin
  - Onkologische Schwerpunktpraxis, Bielefeld
  - Klinikverbund Südwest Kliniken Böblingen Frauenklinik Böblingen, Böblingen
  - Studien GbR Braunschweig, Braunschweig
  - Klinikum Bremen Mitte, Bremen
  - Frauenklinik DIAKO Bremen, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Unifrauenklinik Köln - Studienzentrum Gynäkologie, Cologne
  - St. Elisabeth Hospital, Cologne
  - Kliniken der Stadt Köln / Brustzentrum Holweide, Cologne
  - DONAUISAR Klinikum, Deggendorf
  - Klinikum Dortmund gGmbH, Dortmund
  - St.-Johannes-Hospital Dortmund, Dept. of Obstetrics/Gynecology, Dortmund
  - Onkologische Schwerpunktpraxis, Dresden
  - University Hospital Dresden, Dresden
  - Onkozentrum Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Klinik für Frauenheilkunde & Geburtshilfe, Düsseldorf
  - Frauenklinik der Universität Erlangen, Erlangen
  - Kliniken Essen-Mitte, Klinik für Senologie/ Interdisziplinäres Brustzentrum, Essen
  - Universitätsklinikum Essen, Frauenklinik, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Frankfurt University Department of Gynecology and Obstetrics, Frankfurt
  - AGAPLESION Markus Krankenhaus, Frankfurt am Main
  - Centrum for Haematology and Oncology, Frankurt Am Main
  - Universitätsklinik Freiburg, Klinik für Frauenheilkunde, Freiburg im Breisgau
  - Evangelische Kliniken Gelsenkirchen, Gelsenkirchen
  - MVZ II der Niels-Stensen-Kliniken, Georgsmarienhütte
  - SRH Waldklinikum Gera, Brustzentrum Ostthüringen, Gera
  - MVZ Onkologische Kooperation Harz, Goslar
  - Krankenhaus St. Elisabeth und St. Barbara Halle/Saale, Halle
  - University Medical Center, Hamburg
  - Mammazentrum HH am Krankenhaus Jerusalem, Hamburg
  - Albertinen Krankenhaus, Hamburg
  - Gynäkologisch-Ontologische Praxis Hannover, Hanover
  - DIAKOVERE Henriettenstift Frauenklinik, Hanover
  - Gemeinschaftspraxis Frauenärzte am Bahnhofsplatz, Hildesheim
  - Department of Gyencology and Obstetrics, Saarland University Hospital, Homburg
  - ViDia Christliche Kliniken Karlsruhe, Karlsruhe
  - Elisabethkrankenhaus Kassel, Brustzentrum, Kassel
  - Klinikum Kassel, Kassel
  - University Hospital Schleswig-Holstein, Kiel
  - Institut für Versorgungsforschung in der Onkologie, Koblenz
  - St. Vincenz KH Limburg, Limburg
  - UKSH Campus Lübeck, Lübeck
  - Universitäts-Frauenklinik, Magdeburg
  - Department of Obstetrics and Gynecology, Mainz
  - Medzinische Fakultät Mannheim, Universität Heidelberg, Mannheim
  - Klinikum Memmingen, Memmingen
  - Johannes Wesling Klinikum Minden, Hämatologie-Onkologie/Brustzentrum, Minden
  - Brustzentrum Niederrhein, Mönchengladbach
  - Gynaekologie Arabella, Munich
  - Rotkreuzklinikum München, Frauenklinik, München
  - Medizinisches Versorgungszentrum für Hämatologie und Onkologie München MVZ GmbH, München
  - LMU Klinikum/ Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, München
  - Dept. OB/GYN Johanna Etienne Krankenhaus, Neuss
  - Ortenau Klinikum Offenburg-Kehl, Offenburg
  - Klinikum Oldenburg AöR, Oldenburg
  - Frauenklinik St. Louise - St. Vincenz- Krankenhaus GmbH, Paderborn
  - Klinikum Ernst von Bergmann, Potsdam
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Oncologianova GmbH, Recklinghausen
  - RoMed Klinikum Rosenheim, Rosenheim
  - Univ-Hospital, Dept Ob/Gyn, Rostock
  - CaritasKlinikum St. Theresia, Saarbrücken
  - Onkologische Schwerpunktpraxis Speyer, Speyer
  - G.SUND Gynäkologie Kompetenzzentrum, Stralsund
  - KKH Torgau, Torgau
  - Klinikum Mutterhaus, Trier
  - Praxisnetzwerk Hämatologie/Internistische Onkologie, Troisdorf
  - Frauenklinik, Tübingen
  - Universitätsfrauenklinik Ulm, Ulm
  - Schwarzwald - Baar Klinikum Frauenklinik, Villingen-Schwenningen
  - Harzklinikum Dorothea Christiane Erxleben, Wernigerode
  - St. Anna Hospital Brustzentrum, Witten
  - Klinikum Worms gGmbH, Worms
- Greece (4):
  - General Hospital of Athens Alexandra Clinic, Athens, Attica
  - University General Hospital of Heraklion, Heraklion, Crete
  - University General Hospital of Patras, Pátrai, West Greece
  - General Hospital of Patras Agios Andreas, Pátrai
- Hong Kong (3):
  - Pamela Youde Nethersole Eastern Hospital PYNEH, Hong Kong
  - The Chinese University of Hong Kong (CUHK) - Prince of Wales Hospital (PWH), Hong Kong
  - The University of Hong Kong (HKU) - Queen Mary Hospital (QMH), Pok Fu Lam
- Ireland (5):
  - Saint Vincents University Hospital, Dublin, IE-D
  - St. James Hospital, Dublin, Leinster
  - University College Cork, Cork
  - Mater Misericordiae University Hospital, Dublin
  - University Hospital Limerick, Limerick
- Israel (4):
  - Soroka MC, Beersheba, Southern District
  - Sheba Medical Center, Ramat Gan, Tel Aviv
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Italy (20):
  - Azienda Ospedaliera Garibaldi-Nesima, Catania, CT
  - Istituto Europeo di Oncologia, Milan, MI
  - Clinica Oncologica, Ospedali Riuniti Umberto 1, Ancona
  - Centro di Riferimento Oncologico di Aviano - SOC Oncologia Medica e Prevenzione Oncologica, Aviano
  - Istituto Oncologico di Bari, Bari
  - Azienda ULSS n. 1 Dolomiti, Belluno
  - Policlinico S.Orsola-Malpighi SSD Oncologia Medica Addarii, Bologna
  - SSD Oncologia Medica, Bologna
  - Presidio Ospedaliero di Summa - Antonio Perrino, Brindisi
  - Istituto di Candiolo - IRCCS, Candiolo
  - Ospedale Poli SAN MARTINO, Genova
  - Area Vasta Sud Est Sede Operativa Grosseto, Grosseto
  - Azienda Usl Toscana sud est, Grosseto
  - IRCCS Ospedale San Raffaele, Milan
  - University Hospital of Modena, Modena
  - INT Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - ICS Maugeri IRCCS, Pavia
  - Azienda Ospedaliera di Perugia, Perugia
  - A.O.U. Citta della Salute e della Scienza di Torino, Torino
- Japan (24):
  - Hyogo Cancer Center, Akashi
  - National Cancer Center (NCC) - Tsukiji Campus - National Cancer Center Hospital (NCCH), Chūōku
  - National Hospital Organization - National Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Tokai University Hospital - Isehara Campus, Isehara
  - Sagara Hospital, Kagoshima
  - National Cancer Center Hospital East (NCCHE) - Kashiwa Campus, Kashiwa
  - Japanese Foundation for Cancer Research (JFCR) - The Cancer Institute Hospital - Breast Oncology Center, Kōtoku
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization (NHO) - Shikoku Cancer Center, Matsuyama
  - Aichi Cancer Center Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Hyogo College of Medicine Hospital, Nishinomiya
  - Okayama University Hospital, Okayama
  - National Hospital Organization - Osaka National Hospital (ONH), Osaka
  - Osaka International Cancer Institute (OICI), Osaka
  - Saitama Cancer Center, Saitama
  - National Hospital Organization - Hokkaido Cancer Center, Sapporo
  - Kindai University (Kinki University) - Faculty of Medicine (Kinki University School of Medicine (KUSM)) - Kindai University Hospital (Kinki University Hospital) - Cancer Center, Sayama
  - Tohoku University Hospital (TUH) - Clinical Research, Innovation and Education Center (CRIETO), Sendai
  - Showa University Hospital - Breast Center, Shinagawa-Ku
  - Tokyo Medical University Hospital, Shinjuku-Ku
  - Shizuoka Cancer Center (SCC), Shizuoka
  - Kanagawa Cancer Center Hospital - Kanagawa Cancer Center (Kanagawa Cancer Centre Research Institute), Yokohama
- Mexico (3):
  - CIMAB S.A. de C.V, Torreón, Coahuila
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Consultorio del Dr. Joaqun Gabriel Reinoso Toledo, Monterrey, Nuevo León
- Netherlands (3):
  - Amsterdam UMC - VU Medisch Centrum, Amsterdam, North Holland
  - Amphia Hospital Breda, Breda
  - Erasmus MC - Daniel den Hoed Oncologisch Centrum, Rotterdam
- Peru (4):
  - Hospital Nacional Arzobispo Loayza, Lima
  - Clinica Ricardo Palma, Lima
  - Instituto Nacional de Enfermedades Neoplasicas INEN, Lima
  - Centro de Investigación Clinica Trujillo EIRL, Trujillo
- Poland (5):
  - Centrum Medyczne HCP Sp. z o.o., Poznan, Greater Poland Voivodeship
  - SP Zoz Opolskie Centrum Onkologii IM, Opole, Opole Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - MSCM Cancer Center and Institute of Oncology Department of Breast Cancer and Reconstructive Surgery, Warsaw
- Portugal (10):
  - Hospital da Senhora da Oliveira, Guimarães EPE, Guimarães
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, EPE, Lisbon
  - Fundação Champalimaud, Lisbon
  - Centro Hospitalar de Lisboa Ocidental, EPE, Lisbon
  - Hospital da Luz, Lisbon
  - Hospital CUF Descobertas, Lisbon
  - Hospital Beatriz Ângelo, Loures
  - Unidade Local de Saúde de Matosinhos, EPE, Matosinhos Municipality
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE, Vila Nova de Gaia
- Romania (4):
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca, Cluj
  - Onco Clinic Consult SA, Craiova, Dolj
  - Centrul de Oncologie Sfantu Nectarie, Craiova, Dolj
  - Institutul Oncologic Bucuresti IOB, Bucharest
- Russia (2):
  - SBHI Arkhangelsk Region - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - State Budgetary Healthcare Institution Oncological Dispensary No. 2 of the Ministry of Health of Krasnodar Region, Sochi
- Singapore (2):
  - National University Cancer Institute, Singapore
  - National Cancer Center Singapore, Singapore
- South Korea (11):
  - Kyungpook National University Hospital, Daegu
  - National Cancer Center, Gyeonggi-do
  - CHA Bundang Medical Center CHA University, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center, Irwon-dong
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Songpa-gu
  - Soon Chun Hyang Central Medical Center (SCHMC), Yongsan
- Spain (50):
  - Hospital Universitario de Basurto, Bilbao, Bizkaia
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Sant Joan Reus, Reus, Tarragona
  - Complejo Hospitalario Universitario A Coruña (CHUA), A Coruña
  - Hospital Universitario Fundación Alcorcón, Alcorcón
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de San Juan de Alicante, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital del Mar, Barcelona
  - IOB Institute Of Oncology-Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Mútua Terrassa, Barcelona
  - ALTHAIA, Xarxa Assistencial Universitària de Manresa F.P., Barcelona
  - Hospital de Mataró, Barcelona
  - ICO Hospitalet, Barcelona
  - ICO Badalona, Barcelona
  - Consorcio Hospitalario Provincial de Castelló, Castellon
  - Hospital Universitario San Pedro de Alcantara, Cáceres
  - ICO Girona, Girona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Complejo Hospitalario de Jaen, Jaén
  - Complejo Asistencial Universitario de León, León
  - Hospital Arnau de Vilanova de Lleida, Lleida
  - Clinica Universidad De Navarra, Madrid, Madrid
  - Hospital MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - HM Sanchinarro (CIOCC), Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - Hospital Universitario HM Puerta del Sur, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Rey Juan Carlos, Móstoles
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Hospitalario de Navarra, Navarro
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital General de Catalunya, Sant Cugat del Vallès
  - Complejo Hospitalario Clínico Universitario de Santiago de Compostela (CHUS), Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Quirón Salud Sagrado Corazón, Seville
  - Hospital Universtiario Virgen del Rocio, Seville
  - Fundación Instituto Valenciano de Oncologia (IVO), Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Taiwan (13):
  - E-Da Cancer Hospital, Kaohsiung City, Yanchao District
  - Koo Foundation Sun Yat-Sen Cancer Center, Beitou
  - Changhua Christian Hospital (CCH), Chang-hua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center CMMC - Yongkang Branch, Tainan
  - National Taiwan University Hospital NTUH, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital TPVGH, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital CGMH, Taipei
- Turkey (Türkiye) (4):
  - Hacettepe University Cancer Institute, Ankara, İç Anadolu
  - Trakya University Medical Faculty, Edirne
  - Istanbul Medeniyet University Medical Faculty, Istanbul
  - Medical Park - Izmir Hastanesi, Izmir
- United Kingdom (16):
  - Peterborough City Hospital, Peterborough, Cambridgeshire
  - Kent Oncology Centre Maidstone Hospital, Maidstone, Kent
  - The Christie Hospital, Manchester, Lancashire
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral, Merseyside
  - Nottingham University Hospitals, Nottingham, Nottinghamshire
  - Royal United Hospital Bath NHS Trust - Royal United Hospital RUH, Bath, Somerset
  - Somerset NHS Foundation Trust, Taunton, Somerset
  - St. James University Hospital, Leeds, West Yorkshire
  - Univeristy Hospitals Bristol NHS Foundation Trust, Bristol
  - Colchester Hospital, East Suffolk & North Essex NHS Foundation Trust, Colchester
  - Royal Devon Exeter NHS Foundation Trust, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guys and St Thomas NHS Foundation Trust, London
  - Charing Cross Hospital, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Blackpool Victoria Hospital, Peterborough

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Loibl S, Park YH, Shao Z, Huang CS, Barrios C, Abraham J, Prat A, Niikura N, Im SA, Li W, Li H, Wang Y, Yao H, Kim SB, Geng CZ, Rodriguez Pantigoso W, Ramirez Godinez FJ, Song C, Ching Chang Y, Antoniazzi A, Chen SC, Li Z, Nowecki Z, Lim J, Mathias E, Sato Y, Lu W, Abdel-Monem H, Untch M, Geyer CE Jr; DESTINY-Breast05 Trial Investigators. Trastuzumab Deruxtecan in Residual HER2-Positive Early Breast Cancer. N Engl J Med. 2025 Dec 10. doi: 10.1056/NEJMoa2514661. Online ahead of print. PMID 41370739